CLINICAL TRIAL: NCT04945954
Title: Pharmacokinetic Study of Post-transplant Cyclophosphamide in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Institute of Food and Drug Safety Evaluation (Republic of Korea) (Unknown)
Responsible Party: Principal Investigator, Hyoung Jin Kang, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNUH_MIDD_PTCy
Record Dates: First submitted 2021-06-10; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide (Experimental)
  Interventions: Other: Drug: Cyclophosphamide

INTERVENTIONS:
Other: Drug: Cyclophosphamide — Administer 14.5mg/kg of Cyclophosphamide once a day for 4days. (intravenously)
  Blood sampling of pharmacokinetics(PK) of cyclophosphamide will be performed in all patients who have taken the investigational drug for at least 4 days (For 2 days, It will be administered for pretreatment of transplant, for the other 2 days, It will be administered for Post-transplant treatment for the prevention of GVHD)

SUMMARY:
This is an investigator-initiated clinical trial to analysis population pharmacokinetic characteristics and investigate appropriate pediatric dose of Cyclophosphamide in pediatric hematopoietic stem cell transplantation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had cyclophosphamide treatment for immunosuppressant after allogeneic hematopoietic stem cell transplantation
* Patients age <19 years
* Written Study Informed consent and/or assent from the patient, parent, or guardian

Exclusion Criteria:

* Known hypersensitivity to mycophenolate mofetil or similar class of drug substance
* Patients in a medically critical condition such as severe infection or unstable vital signs
* Any condition that would, in the Investigator's judgment, interfere with full participation in the study
* Subjects who are pregnant or breast-feeding
* Subjects with psychiatric conditions that may interfere with the study
* Subjects who have a possibility of the disease getting worse as a treatment for clinical trials

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameter of melphalan | Day -3: post 2 hour, post 3 hour, post 6 hour, post 24 hour / Day -2: post 2 hour, post 3 hour, post 6 hour( Day 0 means the day when patients receive a HSCT)
  Analysis: Maximum plasma drug concentration (Cmax)
Pharmacokinetics parameter of melphalan | Day +3: post 2 hour, post 3 hour, post 6 hour, post 24 hour / Day +4: post 2 hour, post 3 hour, post 6 hour ( Day 0 means the day when patients receive a HSCT)
  Analysis: Maximum plasma drug concentration (Cmax)
Pharmacokinetics parameter of melphalan | D-3 post 2 hour, post 3 hour, post 6 hour, post 24 hour / D-2 post 2 hour, post 3 hour, post 6 hour / D+3 post 2 hour, post 3 hour, post 6 hour, post 24 hour / D+4 post 2 hour, post 3 hour, post 6 hour( D0 means The day when patients receive a HSCT)
  Analysis: Area under the plasma concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD,PhD, Principal Investigator — l